CLINICAL TRIAL: NCT05728723
Title: The Influence of Android Application as a Pharmaceutical Education Tool on Knowledge, Adherence, Clinical Outcome and Quality of Life of Hypertension Prolanis Patients: A Pilot Study
Brief Title: The Effectiveness of the Android Application as a Pharmaceutical Education Tool in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pharm-202301.01
Record Dates: First submitted 2023-02-05; First posted 2023-02-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
Keywords: Knowledge; Adherence; Quality of Life; Smartphone; Pharmacist
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pharmacy Education with Android Application as a Tool Conducted for Three Months in Hypertensive Patients to Improve Knowledge, Adherence, Outcome Therapy and Quality of Life
  Interventions: Device: Android Application; Behavioral: Pharmacy education
- Pharmacy education (Active Comparator): Pharmacy education in hypertensive patients
  Interventions: Behavioral: Pharmacy education

INTERVENTIONS:
Device: Android Application — Android Application for 3 months
  Arms: Intervention group
Behavioral: Pharmacy education — Pharmacy education in hypertensive patients

SUMMARY:
Hypertension is a worldwide public health challenge due to its high prevalence and along with increased risk of complications of other diseases that are more dangerous if not managed properly. An estimated 1.4 billion people worldwide have high blood pressure, but only 14% can control it. Knowledge of hypertension in patients with hypertension can prevent complications through hypertension treatment. Increasing knowledge can be done by providing education in the form of counseling by pharmacists to hypertensive patients. Counseling activities carried out by pharmacists can be supported by a technological approach. One of the uses in smartphone technology is by creating an android-based mobile application that can be developed to support pharmaceutical care. Education conducted by pharmacists can increase knowledge that will affect hypertension treatment adherence, and this education can also improve blood pressure control so that it can improve the quality of life. The purpose of this study is to analyze the influence of the android application as a standard pharmacist education tool on knowledge as well as adherence and therapeutic outcomes of hypertensive patients, and quality of life related to the health of hypertensive patients compared to just providing standard education by pharmacists to hypertensive patients at the Primary Health Care. The method used in this study is a Quasi-Experimental with Pretest - Posttest Control Group Design. Samples were obtained by purposive sampling method at the selected Primary Health Care as the intervention group and the selected Primary Health Care as the control group. Pharmacist provides education to intervention groups with android applications as counseling aids and in control groups only standard counseling is provided. Pre-test data collection was done by taking primary and secondary data of patients at the first meeting and post-test data collection was taken prospectively through face-to-face interviews and questionnaires on hypertensive patients participants for three months by observing the influence of android applications as counseling aids on knowledge of hypertensive diseases, adherence to antihypertensive treatment, outcome therapy and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years, male and female who are willing to be respondents.
* Patients diagnosed with hypertension or currently taking ≥ 1 antihypertensive drug.
* Hypertension patients who carry out routine control and receive anti-hypertensive drugs for at least 3 months at the Health Center.
* Not illiterate and owns a smartphone.
* Patients who are willing to participate in the study by signing an informed consent.

Exclusion Criteria:

* Physical and mental disabilities such as deaf, blind, and psychiatric disorders.
* The patient is pregnant
* Currently taking hormonal drugs and other routine drugs such as TB, HIV and AIDS drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Knowledge about hypertension | At day 90 after treatment
  Measured by Hypertension Knowledge-Level Scale (HK-LS) questionnaires
Adherence to antihypertensive treatment | At day 90 after treatment
  Measurement by Medication Adherence Report Scale (MARS) questionnaires

SECONDARY OUTCOMES:
Blood pressure | 90 days
  Measurement by blood pressure measuring device.
Quality of life related to the health | 90 days
  Measurement by Short Form-36 (SF-36) questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Abdul K Tasib, S.Si., Apt., Principal Investigator — Faculty of Pharmacy Universitas Padjadjaran Bandung; Eli Halimah, Dr.M.Si.Apt., Principal Investigator — Faculty of Pharmacy Universitas Padjadjaran Bandung; Irma M Puspitasari, Prof.MT.Ph.D, Principal Investigator — Faculty of Pharmacy Universitas Padjadjaran Bandung
Locations (1):
- Health Centers, Bandar Lampung, Lampung, Indonesia